CLINICAL TRIAL: NCT05209815
Title: Safety of Exposure to Natalizumab During Pregnancy
Acronym: BABYZUMAB-2
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2020/65
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Multiple Sclerosis
Keywords: Natalizumab; Safety; pregnancy
MeSH Terms: conditions — Multiple Sclerosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: continuation of NTZ throughout pregnancy and postpartum
  Interventions: Behavioral: Questionnaire
- Group 2: exposure during the first trimester
  Interventions: Behavioral: Questionnaire
- Group 3: exposure during the first and the second trimester
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire

SUMMARY:
Multiple sclerosis (MS) preferentially affects young adults with a female predominance. MS is not associated with an increased risk of complications or abnormal pregnancy outcomes. Nevertheless, disease-modifying therapies can have a teratogenic effect. Discussions about discontinuation should be made with a view to or upon discovery of pregnancy, taking into account the risk of untreated relapses and the risk of toxicity to the fetus.

Natalizumab (NTZ) is a humanized anti-alpha4-integrin monoclonal antibody used as a treatment for highly active relapsing-remitting MS (RRMS). When it is stopped, there is frequent reactivation of the disease with possible relapses and a rebound effect could occur. At present, depending on the center, attitudes of neurologist may vary and 3 main scenarios can be observed: Pregnancy and postpartum under NTZ (group1), Pregnancy partially under NTZ (with or without immunomodulator (IM) supplementation, group 2), or NTZ stopped before pregnancy (with or without IM supplementation, group3).

The first part of the BABYZUMAB study, a retrospective study of Natalizumab exposure during pregnancy, analysed the comparison the clinical activity of the disease (annualized relapse rate) according to these 3 scenarios of NTZ treatment The investigators analyzed the annual relapse rate (ARR) during a two-year period (9 months before and 15 months after the beginning of the pregnancy) in 117 patients identified in the OFSEP database. The investigators showed that the risk of relapses was four times higher in Group 2 versus Group 1 (p=0,014) and six times higher in Group 3 versus Group 1 (p=0,001).

In the literature, there are few studies of newborns from NTZ-exposed pregnancies. No specific pattern of birth defects has been found, but mild to moderate transient thrombocytopenia and anemia have been reported in infants born to NTZ-exposed mothers in the third trimester of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years at the index date (date of pregnancy onset) of data collection,
* RRMS according to McDonald's 2017 criteria (Thompson et al., 2018)
* Affiliated person or beneficiary of a social security scheme.
* followed up at one of the participating centers (OFSEP centers)
* NTZ exposure during pregnancy according to 3 pre-defined sub-groups: continuation of NTZ throughout pregnancy and postpartum (Group 1), exposure during the first trimester (Group 2) exposure during the first and the second trimester (Group 3).
* Participants capable of expressing non objection
* French-speaking, without comprehension disorders

Exclusion Criteria:

* Patient concerned by articles L 1121-5 to L 1121-8 (persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient aged over 18 years old, affected by RRMS according to McDonald's 2017 criteria identified in the BABYZUMAB-1 study
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who presented serious adverse events (SAE) during their pregnancy | At baseline (Day 0)

SECONDARY OUTCOMES:
Proportion of patients who presented pregnancy complications | At baseline (day 0)
Proportion of patients who presented delivery complications | At baseline (day 0)
Proportion of patients who presented postpartum AEs of interest | At baseline (day 0)
Proportion of viable children at birth | At baseline (day 0)
Average weight at birth | At baseline (day 0)
apgar score at birth | At baseline (day 0)
Number of child AEs of interest (haematological, infectious, malformations) at birth | At baseline (day 0)
Number of child AEs of interest (haematological, infectious, malformations) two years after birth | At baseline (day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie RUET, Prof, Principal Investigator — University Hospital, Bordeaux
Locations (27):
- France (26):
  - CHRU de Besançon - service de neurologie, Besançon
  - CHU de Bordeaux - service de neurologie, Bordeaux
  - HCL - service de neurologie, Bron
  - CH Sud Francilien - service de neurologie, Corbeil-Essonnes
  - AP-HP - Hôpital de Créteil - service de neurologie, Créteil
  - CHU de Dijon-Bourgogne, Dijon
  - CHU de Grenoble-Alpes, La Tronche
  - CHRU de Lille - service de neurologie, Lille
  - CHU de Limoges - service de neurologie, Limoges
  - AP-HM - service de neurologie, Marseille
  - CHU de Montpellier - service de neurologie, Montpellier
  - CHRU de Nancy - service de neurologie, Nancy
  - CHU de Nantes - service de neurologie, Nantes
  - CHU de Nice - service de neurologie, Nice
  - CHU de Nîmes - service de neurologie, Nîmes
  - AP-HP - Hôpital La Pitié Salpétrière - service de neurologie, Paris
  - AP-HP - Hôpital Saint-Antoine - service de neurologie, Paris
  - Fondation Rothschild - service de neurologie, Paris
  - CHU de Poitiers - service de neurologie, Poitiers
  - CHU de Rennes - service de neurologie, Rennes
  - CHU de Rouen - service de neurologie, Rouen
  - CH de Saint-Denis - service de neurologie, Saint-Denis
  - CHU d'Amiens - service de neurologie, Salouël
  - CHRU de Strasbourg - service de neurologie, Strasbourg
  - CHU de Toulouse - service de neurologie, Toulouse
  - CHU de Tours - service de neurologie, Tours
- CHU de Fort de France - service de neurologie, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No